CLINICAL TRIAL: NCT03991325
Title: Sonographic Evaluation to Predict Difficult Airway Management
Acronym: US airway
Status: Completed | Type: Observational
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Head of the anesthesia intensive care department, Mongi Slim Hospital
Other Study IDs: sonographic evaluation airway
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Airway Management; Upper Airway Sonographic Evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- difficult laryngoscopy: group of patients with Cormack and Lehane grade III or IV
  Interventions: Diagnostic Test: upper airway sonography
- easy laryngoscopy: group of patients with Cormack and Lehane grade I or II
  Interventions: Diagnostic Test: upper airway sonography

INTERVENTIONS:
Diagnostic Test: upper airway sonography — clinical evaluation of upper airway, ultrasonographic assessement

SUMMARY:
the aim of this study was to evaluate the accuracy of different ultrasonographic parameters and clinical tests to predict difficult airway assessment.

Ultrasonographic parameters were: hyo-mental distence, tongue width, skin to epiglottis distence and skin to hyoid bone distence. these parameters were recorded and their predictive acurracy was studied.

DETAILED DESCRIPTION:
the aim of this study was to evaluate the accuracy of different ultrasonographic parameters and clinical tests to predict difficult airway assessment.

Ultrasonographic parameters were: hyo-mental distence, tongue width, skin to epiglottis distence and skin to hyoid bone distence. these parameters were recorded and their predictive acurracy was studied.

This study analyzed a sample size of 200 patients undergoing elective or urgent surgery under general anesthesia and recieving neuromuscular blocking agent before laryngoscopy.

the correlation between ultrasonographic parameters and difficult laryngoscopy was studied

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for orthopedic or viseral surgery under general anesthesia and tracheal intubation.

Exclusion Criteria:

* patients with suspected tracheal stenosis
* Patients with a poor quality ultrasonographic exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * patients scheduled for orthopedic or viseral surgery under general anesthesia and tracheal intubation.
  Exclusion Criteria:
  * patients with suspected tracheal stenosis
  * Patients with a poor quality ultrasonographic exam
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
prediction of difficult laryngoscopy with ultrasonographic criteria | 5 min after induction of general anesthesia determined by Cormack and Lehane grade
  incidence of difficult laryngoscopy

SECONDARY OUTCOMES:
prediction of difficult mask ventilation with ultrasonographic criteria | 3 min after induction of general anesthesia
  Incidence of difficult ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- Mongi Slim Hospital, La Marsa, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided